CLINICAL TRIAL: NCT05640453
Title: Pregabalin Versus Dexmedetomidine for Delirium Treatment After Coronary Artery Bypass Grafting: A Randomized Double-Blind Trial
Brief Title: Pregabalin Versus Dexmedetomidine for Delirium Treatment After Coronary Artery Bypass Grafting
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Islam Morsy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35912/10/22
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-04

CONDITIONS: Pregabalin; Delirium Treatment; Coronary Artery Bypass Grafting; Dexmedetomidine
MeSH Terms: interventions — Pregabalin; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin group (Active Comparator): Patients will receive pregabalin capsules (75 mg) every 12 h for 24 hours by nasogastric tube.
  Interventions: Drug: Pregabalin
- Dexmedetomidine group (Active Comparator): Patients will receive a bolus dose of 0.4 μg/kg dexmedetomidine (over a period of 10 to 20 min) followed by an infusion of 0.2 to 0.7 μg/h.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Pregabalin — Patients will receive pregabalin capsules (75 mg) every 12 h for 24 hours by nasogastric tube.
  Arms: Pregabalin group
Drug: Dexmedetomidine — Patients will receive a bolus dose of 0.4 μg/kg dexmedetomidine (over a period of 10 to 20 min)
  Arms: Dexmedetomidine group

SUMMARY:
The aim of this study is to determine the effect of pregabalin versus dexmedetomidine on the treatment and lasting duration of delirium in fast tracking elderly patients after Coronary Artery Bypass Grafting.

DETAILED DESCRIPTION:
Delirium is an acute brain disorder that involves changes in consciousness, attention, cognition, and perception.The incidence of postoperative delirium (POD) is high among patients undergoing cardiac surgery, ranging from 20 to 50%, and the risk is even higher in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* CABG patients ≥ 65 years of age both genders American Society of Anesthesiologists (ASA) physical status classification II or III planned for fast track developed postoperative delirium (POD).

Exclusion Criteria:

* Patients who had history of psychiatric diseases; inability to communicate;
* previous history of POD; preoperative sick sinus syndrome, allergy/sensitivity to pregabalin or dexmedetomidine, severe bradycardia (heart rate <50 beat per minute), second-degree or above atrioventricular block without pacemaker; severe hepatic or renal insufficiency.
* Previous cardiac or thoracic surgery, known diagnosis of depression or other major psychiatric diseases, cognitive impairment or inability to cooperate with the study, renal insufficiency, and history of substance abuse.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Percent of delirium treatment | 24 hour postoperatively
  Assessment of delirium will be performed preoperatively and postoperatively at 12-h intervals or as needed according to the patient's condition using the confusion assessment method (CAM)

SECONDARY OUTCOMES:
Level of sedation | 24 hour postoperatively
  Sedation level will be assessed by using the Ramsey sedation scale.
Incidence of weaning from mechanical ventilation | 1 week postoperatively
  percent of patients who weaned from mechanical ventilation
Length of hospital stay | 1 month postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Islam Morsy, Tanta, El-Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will available upon reasonable request from the principal investigator
Supporting Information: Study Protocol, SAP